CLINICAL TRIAL: NCT00654446
Title: A 6-wk Open-Label, Randomised, Multicentre, Phase IIIb, Parallel-Group Study, Which Describes the Renal Effects of the Lipid-Regulating Agents Rosuvastatin and Simvastatin in the Treatment of Sub's With Fredrickson Type IIa & Type IIb Dyslipidaemia, Inc. Heterozygous Familial Hypercholesterolaemia
Brief Title: IIIb 6 Week Open Label Multicentre Rosuvastatin & Simvastatin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Michael Cressman - Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4522IL/0099
Record Dates: First submitted 2008-04-03; First posted 2008-04-08 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Fredrickson Type IIa & Type IIb Dyslipidaemia
Keywords: Cholesterol; low density lipoproteins; dyslipidaemia; Rosuvastatin; Crestor; Simvastatin; Zocor; Renal; kidney
MeSH Terms: conditions — Dyslipidemias | interventions — Rosuvastatin Calcium; Simvastatin

ARMS (2):
- 1 (Experimental): Rosuvastatin
  Interventions: Drug: Rosuvastatin
- 2 (Active Comparator): Simvastatin
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Rosuvastatin
  Other Names: Crestor
  Arms: 1
Drug: Simvastatin
  Other Names: Zocor
  Arms: 2

SUMMARY:
The purpose of this study is to assess the effects on the kidney of rosuvastatin and simvastatin in subjects with Fredrickson Type IIa & Type IIb Dyslipidaemia

ELIGIBILITY:
Inclusion Criteria:

* Fasting low density lipoprotein level as defined by the protocol.
* Fasting triglyceride level as defined by the protocol.

Exclusion Criteria:

* The use of lipid lowering drugs or dietary supplements after Visit 1.
* Active arterial disease eg Unstable angina, or recent arterial surgery
* Blood creatine levels above the limits defined in the protocol or +4 proteinuria during dietary lead in period.
* Uncontrolled hypertension, hypothyroidism, alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442
Dates: Start 2002-09; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Development of Proteinuria | 2 weekly

SECONDARY OUTCOMES:
Renal effects of rosuvastatin and simvastatin | 2 weekly
Low density lipoproteins cholesterol levels | 2 weekly
Safety: adverse events & abnormal laboratory markers | 2 weekly

CONTACTS AND LOCATIONS:
Overall Officials: Evan Stein, Principal Investigator — Metabolic & Athersclerotic research centre, Cincinatti, USA; Russell Esterline, Study Director — AstraZeneca